CLINICAL TRIAL: NCT02280746
Title: Gluten Dietary Intervention for Autistic Symptoms in Children With Autism Spectrum Disorders - Randomized Open Trial
Brief Title: Gluten for Autism Spectrum Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG 8/2013
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - gluten challenge group (Experimental): Gluten challenge group - recommended daily intake of at least one normal meal containing gluten such as bread, pita, pasta, biscuits.
  Interventions: Other: Gluten challenge
- B - gluten-free diet (No Intervention): Continuation of GFD.

INTERVENTIONS:
Other: Gluten challenge — Intervention will be continued for at least 6 months
  Arms: A - gluten challenge group

SUMMARY:
BACKGRUOUND: Autism spectrum disorder (ASD) is a common condition. The etiology of ASD remains unknown. Recent studies suggest a link between elimination diets and severity of autistic symptoms. The possible effects of a gluten-free diet (GFD) on symptoms remain unknown.

AIM: The aim of the study is to evaluate the impact of gluten challenge on the autistic symptoms in children with autism spectrum disorders (ASD) and on a gluten-free diet (GFD) in comparison to individuals continuing GFD.

METHODS: 70 children with ASD aged 3-5 and 11/12 remaining on GFD for at least 8 weeks will be randomly assigned to gluten-free and gluten-challenge diet.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental lifelong disorder, significantly impairing the quality of life of patients and their families. The symptoms are thought to result from interaction between genetics and environment. Treatment is multidisciplinary, based on behavioral therapy, education, and sometimes requires specialized care (i.e. genetics) and pharmacotherapy. The lack of consensus about the etiology of ASD directs researchers to define the condition as combination of symptoms, patient's history data, the impact of co-morbidities (including gastrointestinal disorders), and the effectiveness of various management therapies.

The use of complementary and alternative methods (CAM) of treatment is common and includes especially elimination diets, which are intended to minimize symptoms. The basis for the potentially beneficial impact of dietary intervention has been reported in connection to the correlation between congenital metabolic disorders (phenylketonuria) in patients with ASD and improvements in their overt symptoms in patients with schizophrenia Excessive activity of peptides derived from the metabolism of gluten and casein in individuals with ASD is thought to result in impaired neurotransmission in the brain. The increased permeability of the intestinal barrier, resulting from the inflammatory response (the theory of "leaky gut") in ASD patients, simultaneously promotes excessive absorption of those compounds. Another hypothesis assumes the effectiveness of elimination diets in children with ASD, suggesting allergic background of neuropsychiatric symptoms. Additionally it is emphasized that the lack of ability to communicate symptoms or atypical clinical manifestations (i.e. neuropsychiatric symptoms like hyperactivity, sleep disorders) in children with ASD can make the diagnosis of gastrointestinal symptoms, allergy and other symptoms particularly difficult. Moreover the pain or discomfort may increase the risk of behavioral symptoms.

Review of the literature concerning the effectiveness of gluten-free and casein-free diet (GFCFD) in individuals with ASD reveals a possible bias of the available studies and lack of a definite conclusion. Among 35 identified studies only two randomized controlled trials have been analyzed. The data/information on reported effectiveness of interventions in the behavioral symptoms [mean difference (MD-mean difference) -5.60, 95% CI -9.02 to -2.18, p = 0.001] in Knivsberg's study, is not reliable because of study limitations. Whiteley et al summarized in 2012 the positive effect of GFCFD on various symptoms in ASD patients. However the influence of GFCFD in ASD children can be defined mostly as suggestive because of the methodological limitations. The main biases include: small sample size, unclear process of randomization and allocation, use of different ASD assessment tools, short trial duration, lack of evaluation of patients' compliance to intervention, and other limitations.

The theory of excessive activity of exogenous opioids reports on specific allergies (gluten and casein) suggesting a connection with celiac disease (CD) in subjects with ASD and thus providing a rationale to determine the effect of gluten on gastrointestinal symptoms and consequently on potential behavioral changes in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-5 and 11/12 years with a diagnosis of ASD
* GFD for at least 8 weeks prior to enrollment
* Minimal scores of 15 on SCQ
* Minimal scores 70 points on Leiter scale
* Consent of caregivers to participate in the study

Exclusion Criteria:

* Gluten-mediated disease (celiac disease, wheat allergy)
* Lack of motivation / opportunity to follow a diet
* Malnutrition (defined according World Health Organization - WHO standards as weight for height <-2 SDS - Standard Deviation Scores)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The extent of autistic symptoms based on the Autism Diagnostic Observation Schedule - 2 (ADOS-2) | Change over time - 6 months

SECONDARY OUTCOMES:
The severity of symptoms based on a Social Communication Questionnaire (SCQ) | Change over time - 6 months
Presentation of gastrointestinal (GI) functional disorders (evaluation based on a parent-report form - Rome III diagnostic questionnaire | Before, after 12 weeks and at the end of intervention
The extent of adaptive level of functioning on Vineland Adaptive Behavior Scale (VABS) | Change over time - 6 months
The extent of functioning on Autism Spectrum Rating Scale (ASRS) | Change over time - 6 months
Anthropometry | Change over time - 6 months
  Weight, height based on WHO growth charts, comparison of a ratio of weight for height (WfH), and body mass index (BMI)
Intelligence test Leiter International Performance Scale | Change over time - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Horvath, Study Director — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Piwowarczyk A, Horvath A, Pisula E, Kawa R, Szajewska H. Gluten-Free Diet in Children with Autism Spectrum Disorders: A Randomized, Controlled, Single-Blinded Trial. J Autism Dev Disord. 2020 Feb;50(2):482-490. doi: 10.1007/s10803-019-04266-9. PMID 31659595